CLINICAL TRIAL: NCT03904589
Title: Questionnaires Assessing the Quality of Life of Patients Treated for Coronary Heart Disease: a Pilot Study to Establish Outcome Indicators for Care Pathways From the Patient's Point of View
Brief Title: Questionnaires Assessing the Quality of Life of Patients Treated for Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: José Castro (Other)
Responsible Party: Sponsor-Investigator, José Castro, Head of cardiology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Nyangore
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Heart Disease
  Interventions: Diagnostic Test: Quality of Life assessment

INTERVENTIONS:
Diagnostic Test: Quality of Life assessment — Quality of life will be assessed by means of the Seattle Angina Questionnaire and the Patient Health Questionnaire.

SUMMARY:
Cardiovascular disease remains the leading cause of death in Europe and worldwide. In 2014, they led to more than 4 million deaths in Europe, and coronary heart disease alone accounts for nearly 1.8 million deaths, or 20% of all deaths in Europe. However, mortality from cardiovascular disease and, especially, coronary heart disease has declined in recent decades. This has been made possible by improving the quality of care provided to patients. Several studies have been conducted to demonstrate this improvement in the quality of care, but they mainly measure the functional results of treatment, morbidity and mortality, survival and prolongation of life.

However, patient-centered outcomes such as health-related quality of life outcomes (such as mental function, ability to resume activities of daily living, social relationship) are also considered important outcomes in the management and monitoring of these diseases. Some studies have shown that, even when other risks factors are controlled, a poor quality of life related to health is a prediction factor for morbidity and mortality in patients with coronary artery disease.

Some studies have suggested that health-related quality of life should be strongly associated with lifestyle, co-morbidities, and mental function.

Some factors have been identified as factors that may affect the quality of life in patients with coronary artery disease, including depression, anxiety, dyspnea and angina pectoris. Depression and anxiety were negatively associated with health-related quality of life in patients with cardiovascular disease. As for dyspnea, it has been shown that in stable patients who have had a myocardial infarction, its increase at 1 month after initiation of treatment is strongly associated with a decrease in the quality of life and with an increased risk of re-hospitalization and death. It is therefore important to measure these factors when the quality of life is assessed in patients with coronary heart disease.

The importance of assessing quality of life is that the clinician and the patient often have different concerns: what the clinician considers to be a "successful procedure" is not always considered as such by the patient. Results related to quality of life (results rarely evaluated) are among the results that really interest the patient. Indeed, many patients consider the quality of additional years of life acquired as important as the lifespan, so the goal of today's medicine is to improve the quantity and quality of life of the additional years of life acquired. To ensure this improvement, the assessment of health-related quality of life should be integrated into the daily clinical practice of coronary heart disease management.

The objective of our study is to evaluate the feasibility of this practice throughout the traject of care, by using several standardized questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Confirmed coronary disease

Exclusion Criteria:

Emergencies, patients lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 consecutive patients> 18 years of age admitted to the CHU Brugmann Hospital for coronary artery disease for whom a medical or surgical treatment is considered.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ-7) | Baseline - at hospital admission
  Seattle Angina Questionnaire (SAQ-7), validated and specific questionnaire of angina pectoris which deals with 5 dimensions of quality of life: physical limits, stability of angina, frequency of angina, perception of the disease, satisfaction with the treatment. Each domain has a score calculated on a scale of 0 (= worst health quality) to 100 (= best health quality).
Seattle Angina Questionnaire (SAQ-7) | 1 month after hospital admission
  Seattle Angina Questionnaire (SAQ-7), validated and specific questionnaire of angina pectoris which deals with 5 dimensions of quality of life: physical limits, stability of angina, frequency of angina, perception of the disease, satisfaction with the treatment. Each domain has a score calculated on a scale of 0 (= worst health quality) to 100 (= best health quality).
Seattle Angina Questionnaire (SAQ-7) | 6 months after hospital admission
  Seattle Angina Questionnaire (SAQ-7), validated and specific questionnaire of angina pectoris which deals with 5 dimensions of quality of life: physical limits, stability of angina, frequency of angina, perception of the disease, satisfaction with the treatment. Each domain has a score calculated on a scale of 0 (= worst health quality) to 100 (= best health quality).
Patient Health Questionnaire (PHQ-2) | Baseline - at hospital admission
  Patient Health Questionnaire (PHQ-2) questionnaire used to assess depression. The score is calculated on a scale of 0 (= low possibility of having symptoms related to depression) to 6 (= high possibility of having symptoms related to depression).
Patient Health Questionnaire (PHQ-2) | 1 month after hospital admission
  Patient Health Questionnaire (PHQ-2) questionnaire used to assess depression. The score is calculated on a scale of 0 (= low possibility of having symptoms related to depression) to 6 (= high possibility of having symptoms related to depression).
Patient Health Questionnaire (PHQ-2) | 6 months after hospital admission
  Patient Health Questionnaire (PHQ-2) questionnaire used to assess depression. The score is calculated on a scale of 0 (= low possibility of having symptoms related to depression) to 6 (= high possibility of having symptoms related to depression).

SECONDARY OUTCOMES:
Rose Dyspnea Score | Baseline - at hospital admission
  The Rose Dyspnea Scale is a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Rose Dyspnea Score | 1 month after hospital admission
  The Rose Dyspnea Scale is a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Rose Dyspnea Score | 6 months after hospital admission
  The Rose Dyspnea Scale is a four-item questionnaire that assesses a patients' dyspnea level with common activities. One point is assigned to each activity associated with dyspnea. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea.
Percentage of autonomous filling | 6 months after hospital admission
  Percentage of questionnaires filled autonomously by the patient
Percentage of compliance | 6 months after hospital admission
  Percentage of questionnaires filled by the patient
Average filling time per questionnaire | 6 months after hospital admission
  Average time (in minutes) the patients need to fill one questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Nyangore, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No